CLINICAL TRIAL: NCT03729141
Title: Cholesterol Mobilization and Adipocyte Function in Humans
Brief Title: Dietary Cholesterol and Adipose Tissue Inflammation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study had funding issues and difficulties with recruitment.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00023743
Record Dates: First submitted 2018-10-26; First posted 2018-11-02 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-07

CONDITIONS: Cholesterol
Keywords: Cholesterol; Adipocyte; Macrophage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Added Cholesterol (Experimental)
  Interventions: Dietary Supplement: Added Cholesterol
- No Added Cholesterol (Active Comparator)
  Interventions: Other: No Added Cholesterol

INTERVENTIONS:
Dietary Supplement: Added Cholesterol — Participants assigned to the added cholesterol group will receive snacks containing added cholesterol (1g/day) for 3 weeks prior to surgery.
  Arms: Added Cholesterol
Other: No Added Cholesterol — Participants assigned to the no added cholesterol group will receive snacks containing no added cholesterol for 3 weeks prior to surgery.
  Arms: No Added Cholesterol

SUMMARY:
Hypothesis: increasing dietary cholesterol in humans will increase visceral, but not subcutaneous adipocyte size, free cholesterol content, and inflammatory gene expression.

Visceral and abdominal subcutaneous adipose tissue biopsies will be obtained from non-obese subjects undergoing elective abdominal surgery at Wake Forest Baptist Medical Center after 3 weeks of zero (control) or 1g dietary cholesterol supplementation. Blood samples will also be taken before and after 3 weeks of dietary supplementation (0 vs. 1g dietary cholesterol) to measure plasma lipids levels, and ex vivo monocyte chemotaxis. Blood will also be used to isolate CD14+ monocytes for RNA extraction and storage for future transcriptome studies. Measurements of adipocyte size, free cholesterol content, and inflammatory gene and protein expression in the adipose tissue biopsies to test the hypothesis. Adipocytes and the stromal vascular fraction will be isolated and evaluated for CD14+ macrophages for RNA extraction and storage for future transcriptome analysis.

DETAILED DESCRIPTION:
A Wake Forest School of Medicine Clinical Research Unit-based pilot study will be conducted in which subjects scheduled to undergo elective intra-abdominal surgery at Wake Forest Baptist Medical Center (i.e., cholecystectomy, Nissen fundoplication, hernia repair, etc.) will be recruited. Subjects will be randomly and blindly assigned to receive daily treats (cookie, brownie, or muffin) containing either no added cholesterol (control) or 1g of cholesterol/day (~0.4 mg/Kcal cholesterol) for 3 weeks prior to surgery. Three weeks for the length of cholesterol supplementation has been chosen because this is within the duration of human egg-consumption studies in which significant elevations in plasma LDL concentrations occurred. A blood sample will be taken from each participant at baseline before starting the supplementation period and after 3 weeks of 0 or 1g/day cholesterol supplementation, at the time of scheduled surgery. The blood samples will be used for measurement of lipid profile, ex vivo monocyte chemotaxis, and for monocyte RNA isolation. During surgery, abdominal wall subcutaneous adipose tissue and mesenteric (visceral) adipose tissue samples will be obtained. Aliquots of adipose tissue will be fixed overnight for histology and measurement of adipocyte size distribution and CD68 immunostaining, flash frozen and stored for cholesterol quantification by gas liquid chromatography, extracted to isolate RNA and protein for quantitative real time PCR and immunoblotting of inflammatory gene and protein expression, and collagenase digested to isolate adipocytes and stromal vascular cell fraction macrophages which will be used to extract and store RNA for future transcriptome analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age:18 to 70 years old
* Operated on by one of the study team surgeons at Wake Forest Baptist Medical Center.

Exclusion Criteria:

* History of liver disease (e.g., autoimmune hepatitis, Wilson's disease, hemochromatosis, 1 anti-trypsin deficiency), as determined by chart review
* Childs A, B, or C cirrhosis, as determined by chart review
* Present diagnosis/treatment of malignancy other than non-melanoma skin cancer
* Baseline INR > 1.8, as determined by chart review or need for continuous anticoagulation with warfarin or heparin
* Platelets <50,000 as determined by chart review
* Active immunomodulation therapy for chronic inflammatory diseases, including but not limited to rheumatoid arthritis, psoriasis, SLE, sarcoidosis, or inflammatory bowel disease
* Diabetes mellitus requiring treatment with oral agents or insulin
* Taking Questran, Colestid, or Zetia
* BMI over 30

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Plasma total | up to 6 weeks after surgery
  Plasma will be used to measure plasma total
Adipocyte size | within 6 weeks after surgery
  Adipocyte size will be evaluated by histology by microscopic examination and morphometry.
Lipoprotein cholesterol levels | up to 6 weeks after surgery
  Plasma will be used to measure lipoprotein cholesterol levels.

OTHER OUTCOMES:
Plasma lipid levels | up to 12 weeks
  Blood samples will be collected from subjects at baseline and at the time of surgery in which snacks containing either no added cholesterol or 1g/day added cholesterol were eaten for three weeks prior to surgery. Plasma lipid levels will be measured. In addition blood will be used to isolate CD14+ monocytes for RNA extraction and storage for future transcriptome studies.
Ex vivo monocyte chemotaxis | up to 12 weeks
  Blood samples will be collected from subjects at baseline and at the time of surgery in which snacks containing either no added cholesterol or 1g/day added cholesterol were eaten for three weeks prior to surgery. Ex vivo monocyte chemotaxis will be measured. In addition blood will be used to isolate CD14+ monocytes for RNA extraction and storage for future transcriptome studies.
Gene expression | within 20 weeks of surgery.
  Visceral and subcutaneous adipose tissue will be collected from subjects in which snacks containing either no added cholesterol or 1g/day added cholesterol were eaten for three weeks prior to surgery. Tissue samples will be taken from non-obese participants undergoing elective abdominal surgery to be used to measure inflammatory gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Weinberg, MD, Principal Investigator — Wake Forest University Health Sciences; John Parks, Ph.D, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States